CLINICAL TRIAL: NCT00658086
Title: A Multi-Center, Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Safety and Antiviral Activity of Aerosolized ALN-RSV01 Plus Standard of Care in Lung Transplant Patients Infected With Respiratory Syncytial Virus (RSV)
Brief Title: Phase 2 Study of ALN-RSV01 in Lung Transplant Patients Infected With Respiratory Syncytial Virus (RSV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Jared Gollob, MD Sr. Director Clinical Research, Alnylam Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-RSV01-106
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: ALN-RSV01; Respiratory Syncytial Virus
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): ALN-RSV01
  Interventions: Drug: ALN-RSV01
- 2 (Placebo Comparator): Normal saline
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: ALN-RSV01 — administered by nebulization once daily for 3 days
  Arms: 1
Drug: normal saline — administered by nebulization once daily for 3 days
  Arms: 2

SUMMARY:
To evaluate the safety,tolerability and antiviral activitity of ALN-RSV01 in RSV infected lung transplant patients

ELIGIBILITY:
Inclusion Criteria:

* Single or bilateral lung transplant recipients
* Confirmed RSV infection
* Greater than 90 days post current lung transplant
* Rejection free for a minimum of 1 month

Exclusion Criteria:

* Antimicrobial therapy for known viral, bacterial, or fungal respiratory co-infection at the time of diagnosis
* Bronchiolitis obliterans syndrome (BOS) Grade 3 or any state BOS with FEV1 that has not been stable for at least 3 months
* Use of alemtuzumab within 9 months prior to screening; anti-thymocyte globulin(ATG) or thymoglobulin within 3 months of screening: concurrent use of >= 0.3 mg/kg/day prednisone or equivalent as maintenance therapy
* active treament for acute graft rejection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Assess safety and tolerability of aerosolized ALN-RSV01 versus placebo in lung transplant patients infected with RSV | Day 30

SECONDARY OUTCOMES:
Evaluate effects of ALN-RSV01 on clinical and virologic endpoints | Throughout Trial

CONTACTS AND LOCATIONS:
Overall Officials: Martin Zamora, MD, Principal Investigator — University of Colorado Health Science Center; Allan Glanville, MB BS MD Syd, FRACP, Principal Investigator — St. Vincent's Hospital NSW Australia
Locations (13):
- United States (10):
  - Clinical Site, San Diego, California
  - Clinical Site, San Francisco, California
  - Clinical Site, Denver, Colorado
  - Clinical Site, Gainesville, Florida
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Chicago, Illinois
  - Clinical Site, Boston, Massachusetts
  - Clinical Site, Minneapolis, Minnesota
  - Clinical Site, Cleveland, Ohio
  - Clinical Site, Nashville, Tennessee
- Australia (3):
  - Clinical Site, Sydney, New South Wales
  - Clinical Site, Brisbane, Queensland
  - Clinical Site, Perth, Western Australia

REFERENCES:
- [Derived] Zamora MR, Budev M, Rolfe M, Gottlieb J, Humar A, Devincenzo J, Vaishnaw A, Cehelsky J, Albert G, Nochur S, Gollob JA, Glanville AR. RNA interference therapy in lung transplant patients infected with respiratory syncytial virus. Am J Respir Crit Care Med. 2011 Feb 15;183(4):531-8. doi: 10.1164/rccm.201003-0422OC. Epub 2010 Sep 17. PMID 20851929